CLINICAL TRIAL: NCT01901679
Title: A Pilot Study: Celecoxib Inhibition of Aromatase Expression and Inflammation in Adipose Tissue of Obese Postmenopausal Women
Brief Title: Celecoxib Inhibition of Aromatase Expression and Inflammation in Adipose Tissue of Obese Postmenopausal Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHO-0807
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity; Post-menopausal
MeSH Terms: conditions — Obesity | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celebrex (Experimental): 10 days treatment with Celebrex to evaluate reduction of PGE-M in urine
  Interventions: Drug: Celebrex

INTERVENTIONS:
Drug: Celebrex — 200 mg PO BID
  Other Names: Celecoxib

SUMMARY:
The study plans to find out whether Celebrex may be potentially useful to decrease inflammation in fat tissues and thereby lower the production of substances such as estrogens that may increase the risk of developing breast cancer and lead to a poor outcome of the disease.

DETAILED DESCRIPTION:
This study seeks to examine how effective the celebrex may be in reducing inflammation, crown-like structures in fat tissue, the enzyme aromatase, PGE-M in the urine and estrogen in blood and urine. Volunteer subjects will be expected to stay in the hospital for about 2 weeks taking Celebrex for approximately 10 days while eating a diet similar to what they consumed before coming into the hospital for the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman defined as: 24 consecutive months without a menstrual period and currently not taking any medication known to induce amenorrhea.
* Serum estradiol < 20 pg/mL
* Body Mass Index of 35-50
* Stable weight defined as (+/- 5 %) of body weight for at least three months
* 40-70 years of age
* Fluent in English

Exclusion Criteria:

* Known hypersensitivity to celecoxib or sulfonamides
* Known peptic ulcer disease
* Hypertension BP > 150/90 (on 2 occasions after resting)
* Fasting blood glucose > 165 mg/dL
* HIV positive
* Screening creatinine > 2X upper limit of normal
* Screening LFT results > 2x upper limit of normal
* Smokers (or stopped < 3 months ago)
* Framingham risk score > 15
* Evidence of active coronary disease by history and/or EKG
* Subjects who consume 25 grams of soy protein/day or more than 45 mg of isoflavones/day, for subjects who consume this amount of soy, they may stop for 14 days prior to admission
* Currently taking NSAIDS, aspirin, (if > once a week, stopped <30 days ago).
* Consuming > 3 servings of fish or seafood/week
* Currently taking fish oil, omega-3 supplements or other herbal supplements that exceed GRAS (Generally Recognized as Safe) levels, (if currently taking fish oil/omega-3 supplements, there must be a 30 day washout period)
* Current use of anti-coagulants
* Currently taking any weight control medication
* Currently taking thioridazine
* Currently taking lithium
* Currently taking any estrogen/progesterone hormones including vaginal cream, e-string, or vaginal tablets
* Currently taking any medication that can alter fat stores as determined by the principal investigator
* History of Inflammatory Bowel Disease or other chronic inflammatory disorders
* History of any malignancy other than non-melanoma skin cancer in the past 5 years
* History of any bleeding disorder
* History of cardiovascular disease
* Diagnosis of asthma
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted during 2 outpatient visits at Rockefeller University Hospital outpatient clinic. Recruitment of subjects began on 6/10/13 and was completed on 6/30/14.
Pre-assignment Details: All participants were screened for their usual dietary intake and instructed to continue to follow their usual diet during weeks prior to hospital admission and thoughout the entire study. .
  First group underwent 3 day run-in period inpatient, the second group underwent 14 day run-in period prior to starting Celecoxib 200mg po BID X 10 days.
Groups:
- 1st Group: 3 Day run-in Period: After 3 day run-in period, participants underwent baseline testing then started 10 days of Celecoxib 200mg po BID. Follow-up blood and stool collection was performed as outpatients 7-10 days after discharge.
- 2nd Group: 14 Day run-in Period: After 14 day run-in period, participants underwent baseline testing then started 10 days of Celecoxib 200mg po BID. Follow-up blood and stool collection was performed as outpatients 7-10 days after discharge.
Period: Overall Study
Arm/Group | 1st Group: 3 Day run-in Period | 2nd Group: 14 Day run-in Period
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3 Day run-in Period: After 3 day run-in period, participants underwent baseline testing then started 10 days of Celecoxib 200mg po BID. Follow-up blood and stool collection was performed as outpatients 7-10 days after discharge.
- 14 Day run-in Period: After 14 day run-in period, participants underwent baseline testing then started 10 days of Celecoxib 200mg po BID. Follow-up blood and stool collection was performed as outpatients 7-10 days after discharge.
- Total: Total of all reporting groups
Arm/Group | 3 Day run-in Period | 14 Day run-in Period | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 62 [56 to 68] | 56 [53 to 60] | 59 [53 to 68]
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
BMI [Mean (Full Range); unit: kg/m^2] | 40.2 [38.2 to 43.1] | 39.7 [36.7 to 45.1] | 40.0 [36.7 to 45.1]

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether Oral Administration of Celebrex to Obese Women Will Reduce the PGE-M in Urine
Description: Study endpoint is a reduction in PGE-M in urine after treatment with celebrex
Time Frame: 10 days
Population: These samples were collected but not analyzed due to technical reasons. Investigator has retired and access to results was not available for this outcome. Best efforts were made to obtain the data; however, they were unsuccessful.
Arm/Group | 1st Group: 3 Day run-in Period | 2nd Group: 14 Day run-in Period
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Collected during inpatient phase of study, an average of 14 days for 3 day run-in period or 24 days for 14 day run-in period
Description: AE's were reported when discovered. Reports were from investigator assessment, nursing assessment and patient complaints. All AE's were documented and submitted to the IRBand PI as per protocol.
Arm/Group | 1st Group: 3 Day run-in Period | 2nd Group: 14 Day run-in Period
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1st Group: 3 Day run-in Period (N=5) | 2nd Group: 14 Day run-in Period (N=5)
hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — During abdominal fat biopsy procedure, there was moderate bleeding from the site. Procedure was stopped, and the bleeding ceased. Subject was stable and recovered promptly, but was monitored for an additional day for safety.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1st Group: 3 Day run-in Period (N=5) | 2nd Group: 14 Day run-in Period (N=5)
bruise at biopsy site (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) — Due to the pinching of abdominal fat during the fat biopsy, a resultant bruise medial to the incision is common and expected. It resolved within 3-4 days and well tolerated. The risk is addressed in the informed consent.
burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant spilled hot tea on her chest wall resulting in 1st degree scald burn of her upper chest.
atypical chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Subject complained of chest pain after burning her skin with hot tea.
elevated serum cholesterol (Investigations) | 0 (0) | 1 (1) — Subjet had history of hypercholesteremia. She stopped taking statin medication prescribed by PMD. Cholesterol level increased. PMD was informed and given test results.
elevated ALT (Investigations) | 0 (0) | 1 (1) — After 10 days on celecoxib, subject had mild elevation in ALT
GI Bloating and constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject complained of bloating and constipation.
sore throat and dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject complained of sore throat and dry cough after a group gathering. Afebrile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT01901679/Prot_SAP_000.pdf